CLINICAL TRIAL: NCT00818805
Title: Efficacy Investigation Study of Olopatadine Hydrochloride Ophthalmic Solution Using OHIO Chamber in Patients With Seasonal Allergic Rhinitis (SAR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AL-292ET
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2010-03-15 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2010-03

CONDITIONS: Allergic Conjunctivitis
Keywords: conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic; Conjunctivitis | interventions — Olopatadine Hydrochloride; tranilast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Olopatadine 0.1% one eye (Experimental): Patients received one drop Olopatadine 0.1% in one eye and 1 drop Olopatadine placebo in contralateral eye
  Interventions: Drug: Olopatadine 0.1%
- Tranilast 0.5% one eye (Experimental): Patients received one drop Tranilast ophthalmic solution 0.5% in one eye and 1 drop tranilast placebo in contralateral eye
  Interventions: Drug: Tranilast 0.5%
- Placebo (Olopatadine) (Placebo Comparator): Patients received one drop Olopatadine 0.1% in one eye and 1 drop Olopatadine placebo in contralateral eye
  Interventions: Drug: Placebo (Olopatadine)
- Placebo (Tranilast) (Placebo Comparator): Patients received one drop Tranilast ophthalmic solution 0.5% in one eye and 1 drop tranilast placebo in contralateral eye
  Interventions: Drug: Placebo (Tranilast)

INTERVENTIONS:
Drug: Olopatadine 0.1% — one drop in one eye
  Arms: Olopatadine 0.1% one eye
Drug: Tranilast 0.5% — one drop in one eye
  Arms: Tranilast 0.5% one eye
Drug: Placebo (Olopatadine) — one drop in contralateral eye
  Arms: Placebo (Olopatadine)
Drug: Placebo (Tranilast) — one drop in contralateral eye
  Arms: Placebo (Tranilast)

SUMMARY:
To evaluate the efficacy of olopatadine 0.1% using the OHIO Chamber in patients with seasonal allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age/Gender: males and females aged >20 to < 65 years (at the time of obtaining consent).
2. Positive cases in whom blood specific IgE antibody quantification against cedar pollen showed class 2-6 in a health checkup conducted within the past 3 years.
3. Cases who were diagnosed as patients with seasonal allergic conjunctivitis and were judged eligible as subjects of the said study by the investigator or co-investigator from the results of medical examination conducted on the day of the study or prior to it.
4. Cases who gave consent on study participation of their own free will in writing, with understanding the contents of the said study.

Exclusion Criteria:

1. Cases with an ocular disease that requires treatment other than allergic conjunctivitis.
2. Cases with an inflammatory ocular disease in the external/anterior part of the eye that may affect drug efficacy evaluation.
3. Cases with a respiratory disease such as bronchial asthma other than allergic rhinitis.
4. Cases with past history of anaphylaxis.
5. Cases with past history of hypersensitivity to olopatadine hydrochloride/tranilast.
6. Cases undergoing immunotherapy (hyposensitization therapy; modulated therapy).
7. Patients who are pregnant, lactating women, or may be pregnant, or cases wishing to be pregnant during the study period.
8. Other cases who are judged ineligible for participation in the main study by the doctor in charge of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period: May 21-31, 2008 Location: Samoncho Clinic
Pre-assignment Details: The study was conducted using an Ohio chamber in two parts: 1) a proof-of concept pilot study designed to assess the appropriateness of the OHIO chamber to induce ocular symptoms. 2) a randomized, single-masked, placebo-controlled, cross-over study.
Groups:
- Olopatadine 0.1% First, Then Tranilast Second: Patients received Olopatadine 0.1% one eye/ Placebo (Olopatadine) in contralateral eye first, then received Tranilast 0.5% one eye/ Placebo (Tranilast) in contralateral eye next
- Tranilast 0.5% First, Then Olopatadine Second: Patients received Tranilast 0.5% one eye/ Placebo (Tranilast) in contralateral eye first, then received Olopatadine 0.1% one eye/ Placebo (Olopatadine) in contralateral eye last.
Period: First Intervention
Arm/Group | Olopatadine 0.1% First, Then Tranilast Second | Tranilast 0.5% First, Then Olopatadine Second
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Olopatadine 0.1% First, Then Tranilast Second | Tranilast 0.5% First, Then Olopatadine Second
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in "Ocular Itching" Score (5-point Scale) in Subjective Symptom Questionnaire
Description: Ocular itching score was assessed using a 5 point scale, with 1 meaning no itching and 4 meaning worst itching.
Time Frame: 0-180 minutes after entering the examination room
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Olopatadine 0.1% One Eye: Olopatadine 0.1% in one eye in either the first or second period
- Tranilast 0.5% One Eye: Tranilast 0.5% in one eye in either the first or second period
- Placebo (Olopatadine): Placebo (Olopatadine) in one eye in either the first or second period
- Placebo (Tranilast): Placebo (Tranilast) in one eye in either the first or second period
Arm/Group | Olopatadine 0.1% One Eye | Tranilast 0.5% One Eye | Placebo (Olopatadine) | Placebo (Tranilast)
Number analyzed (Participants) | 50 | 50 | 50 | 50
Units on a scale
  15 minutes | 0.19 (0.47) | 0.11 (0.46) | 0.06 (0.33) | 0.08 (0.44)
  30 minutes | 0.44 (0.61) | 0.25 (0.50) | 0.33 (0.53) | 0.28 (0.51)
  45 minutes | 0.50 (0.70) | 0.36 (0.68) | 0.50 (0.65) | 0.56 (0.69)
  60 minutes | 0.67 (0.76) | 0.50 (0.74) | 0.75 (0.69) | 0.61 (0.73)
  75 minutes | 0.81 (0.82) | 0.67 (0.79) | 0.92 (0.81) | 0.78 (0.76)
  90 minutes | 0.92 (0.81) | 0.86 (0.72) | 0.92 (0.69) | 0.94 (0.75)
  105 minutes | 0.94 (0.58) | 0.86 (0.72) | 1.03 (0.70) | 0.97 (0.81)
  120 minutes | 1.03 (0.65) | 1.03 (0.70) | 1.19 (0.67) | 1.08 (0.81)
  135 minutes | 1.17 (0.70) | 1.14 (0.72) | 1.33 (0.72) | 1.19 (0.82)
  150 minutes | 1.25 (0.77) | 1.14 (0.76) | 1.36 (0.64) | 1.25 (0.77)
  165 minutes | 1.28 (0.78) | 1.14 (0.76) | 1.39 (0.64) | 1.33 (0.76)
  180 minutes | 1.39 (0.77) | 1.39 (0.77) | 1.44 (0.69) | 1.47 (0.88)

2. Secondary Outcome: Change in Total Score in Ocular Symptom Questionnaire
Time Frame: 15-180 min.
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Placebo (Olopatadine) One Eye: Placebo (Olopatadine) in one eye in either the first or second period
- Placebo (Tranilast) One Eye: Placebo (Tranilast) in one eye in either the first or second period
Arm/Group | Olopatadine 0.1% One Eye | Tranilast 0.5% One Eye | Placebo (Olopatadine) One Eye | Placebo (Tranilast) One Eye
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No